CLINICAL TRIAL: NCT04573803
Title: Pharmacological Management of Seizures Post Traumatic Brain Injury (MAST)
Brief Title: Pharmacological Management of Seizures Post Traumatic Brain Injury
Acronym: MAST
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Peter Hutchinson, Professor of Neurosurgery & Honorary Consultant Neurosurgeon, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A095460
Record Dates: First submitted 2020-09-07; First posted 2020-10-05 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury; Post Traumatic Seizures
Keywords: Phenytoin; Levetiracetam; Post-traumatic seizure; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Phenytoin; Levetiracetam

STUDY DESIGN:
Intervention Model Description: The MAST trial consists of two pragmatic, open-label, multi-centre, independent, parallel, randomised trials. MAST-DURATION consists of two arms and MAST-PROPHYLAXIS consists of three arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MAST DURATION - <3 months (Experimental): TBI patients with early seizures (within first 7 days following trauma) will receive a short course of up to 3 months of either Phenytoin Sodium or Levetiracetam.
  Interventions: Drug: Phenytoin Sodium; Drug: Levetiracetam
- MAST DURATION - >6 months (Experimental): TBI patients with early seizures (within first 7 days following trauma) will receive a longer course of at least 6 months of either Phenytoin Sodium or Levetiracetam.
  Interventions: Drug: Phenytoin Sodium; Drug: Levetiracetam
- MAST PROPHYLAXIS - Phenytoin Sodium (Experimental): TBI patients, without an acute symptomatic seizure, will receive a 7-day course of Phenytoin Sodium as seizure prophylaxis.
  Interventions: Drug: Phenytoin Sodium
- MAST PROPHYLAXIS - Levetiracetam (Experimental): TBI patients, without an acute symptomatic seizure, will receive a 7-day course of Levetiracetam as seizure prophylaxis. Dosing will be as prescribed clinically by the treating physician.
  Interventions: Drug: Levetiracetam
- MAST PROPHYLAXIS - no treatment (No Intervention): TBI patients, without an acute symptomatic seizure, will not receive any anti-epileptic drug.

INTERVENTIONS:
Drug: Phenytoin Sodium — Dosing will be as prescribed clinically by the treating physician. Phenytoin Sodium may be administered orally, intravenously or via nasogastric tube.
  Arms: MAST DURATION - <3 months; MAST DURATION - >6 months; MAST PROPHYLAXIS - Phenytoin Sodium
Drug: Levetiracetam — Dosing will be as prescribed clinically by the treating physician.Levetiracetam may be administered orally, intravenously or via nasogastric tube.
  Other Names: Keppra
  Arms: MAST DURATION - <3 months; MAST DURATION - >6 months; MAST PROPHYLAXIS - Levetiracetam

SUMMARY:
The overall aim of the MAST trial is to define best practice in the use of anti-epileptic drugs (AEDs) for patients following a traumatic brain injury (TBI). The trial will consist of two parts. The first part aims to answer whether a shorter or a longer course of AEDs is better to prevent further seizures in patients who have started having seizures following TBI (MAST - duration). The second part aims to answer whether a 7-day course of either Phenytoin or Levetiracetam should be used for patients with a serious TBI to prevent seizures from starting (MAST- prophylaxis).

DETAILED DESCRIPTION:
The majority of patients who suffer a traumatic brain injury (TBI) do not need to stay in hospital overnight. However, some require admission to a specialist hospital, as their injury is more serious. Seizures can be harmful or even fatal, if not treated appropriately. Medications that reduce the risk of seizures are called antiepileptic drugs (AEDs). However, AEDs have side effects, which can affect patients' quality of life, memory, concentration and general health.

Patients with seizures after TBI are typically prescribed an AED to prevent further seizures, most commonly Phenytoin or Levetiracetam. Some doctors favour a short course, whereas others favour a longer course. The first part of the trial aims to answer if one approach is better than the other (MAST-duration). The second part of the trial aims to answer if a 7-day course of either Phenytoin or Levetiracetam should be used for patients with a serious TBI to prevent seizures from happening (MAST- prophylaxis).

All patients admitted to a neurosurgical unit (NSU) within the UK, with a serious TBI, will be considered for the trial. Patients who have been started on either Phenytoin or Levetiracteam by their clinical team due to seizures will be randomised to either up to 3 months or at least 6 months of treatment. In an independent, parallel trial, TBI patients who have not had a seizure will be randomised to phenytoin, levetiracetam or no treatment. All patients will be managed as per usual NHS practice and followed up for 24 months.

ELIGIBILITY:
MAST DURATION

Inclusion Criteria:

* Patients aged ≥10 years with TBI managed in an NSU who have started on an phenytoin or levetiracetam due to an acute symptomatic seizure during acute hospitalisation
* Patient or Legal Representative is willing and able to provide informed consent or in the absence of a legal representative, an Independent Healthcare Professional provides authorisation for patient enrolment

Exclusion Criteria:

* Unsurvivable injury
* Previous history of epilepsy
* Patients who are on an AED pre-TBI
* Patient who has been clinically prescribed an AED other than phenytoin or levetiracetam
* Unwillingness to take products containing gelatin (animal products)
* Severe lactose intolerance or any known hypersensitivity to study drug or any of its excipients

MAST-PROPHYLAXIS

Inclusion Criteria:

* Patients aged ≥10 years, with TBI managed in an NSU without an acute symptomatic seizure
* Patient or Legal Representative is willing and able to provide informed consent or in the absence of a legal representative, an Independent Healthcare Professional provides authorisation for patient enrolment within 48 hours of admittance.

Exclusion Criteria:

* Post-traumatic seizures
* Unsurvivable injury
* Previous history of epilepsy
* Patients who are on an AED pre-TBI
* Pregnancy or breastfeeding
* Unwillingness to take products containing gelatin (animal products)
* Severe lactose intolerance or any known hypersensitivity to study drug or any of its excipients
* Time interval from the time of admission to NSU to randomisation exceeds 48 hours

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1649 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
MAST-DURATION: Occurrence of late PTS | Within 24 months post traumatic brain injury
  The primary outcome for MAST-DURATION is the occurrence of late post-traumatic seizure. This will be assessed by follow-up questionnaire.
MAST-PROPHYLAXIS: Occurrence of PTS | Within 2 weeks post TBI
  The primary outcome for MAST-PROPHYLAXIS is the occurrence of an acute symptomatic seizure. This will be assessed in the neurosurgical unit, or by telephone following discharge.

SECONDARY OUTCOMES:
MAST-PROPHYLAXIS: Occurrence of post-traumatic seizures | Within 24 months post traumatic brain injury
  The occurrence of post-traumatic seizures. This will be assessed by follow-up questionnaire.
MAST-PROPHYLAXIS: Time to post-traumatic seizure | Within 24 months post traumatic brain injury
  The time to post traumatic seizure. This will be assessed by follow-up questionnaire.
Both trials: Disability | At 6, 12, 18 and 24 months
  Levels of disability will be assessed using the Extended Glasgow Outcome Scale via follow-up questionnaire. The scale is scored from 1 (death) to 8 (upper good recovery) with higher scores reflecting a better outcome.
Both trials: Cognitive function | At 6, 12, 18 and 24 months
  Cognitive function will be assessed using the Neurobehavioural Symptom Inventory via follow-up questionnaire. Symptoms are scored from 0 (mild) to 4 (very severe) with higher scores reflecting a worse outcome.
Both trials: Quality of life | At 6, 12, 18 and 24 months
  Quality of life will be assessed using the EQ-5D-5L via follow-up questionnaire. The EQ-5D-5L consists of 2 parts - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale. The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) which are scored from 1 (no problems) to 5 (extreme problems) with higher scores reflecting a worse outcome. The EQ Visual Analogue scale is numbered 0 to 100 with higher scores reflecting a better outcome.
Both trials: Adverse events | At 6, 12, 18 and 24 months
  Adverse events will be assessed using the Liverpool Adverse Events Profile via follow-up questionnaire. The questionnaire is scored from 1 (never a problem) to 4 (always or often a problem) with higher scores reflecting a worse outcome.
Both trials: Hospital admissions | Within 24 months post traumatic brain injury
  Hospital admissions will be extracted from the NHS Digital Hospital Episode Statistics (HES) database) and equivalents. Hospital admissions will be combined with the length of anti-epileptic drug treatment to report an economic evaluation.
Both trials: Frequency of PTS | Within 24 months post traumatic brain injury
  The frequency of post traumatic seizures.
Both trials: Mortality | At 6, 12, 18 and 24 months
  Death from any cause
Both trials: Frequency of adverse events of special interest | Up to 24 months
  Frequency of adverse events of special interest (unfavourable and unintended sign, symptom, or disease temporally associated with the use of trial drug, whether or not considered related to the trial drug.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hutchinson, PhD, Principal Investigator — University of Cambridge